CLINICAL TRIAL: NCT01287273
Title: The Impact of Early Embryos Incubation on Pregnancy Rate in IVF
Acronym: IVF-2010
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Martha Dirnfeld (Other)
Responsible Party: Sponsor-Investigator, Martha Dirnfeld, Head of IVF Unit, Carmel Medical Center
Organization: Carmel Medical Center (Other)
Other Study IDs: CMC-10-0010-CTIL
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy; In Vitro Fertilization
Keywords: frozen-thawed; IVF; incubation; pregnancy rate; Pregnancy rate of frozen-thawed embryos of IVF treatments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Transfer at the day of embryo thawing
- Group B: Transfer of thawed embryos 24-72 hours post thawing

SUMMARY:
Frozen- thawed embryos obtained by IVF treatments are transferred to the uterus immediately following thawing or after incubation for additional 24-72 hours. The two methods are routine in IVF laboratories. In this study the investigators would like to compare between these two methods in terms of implantation rate, pregnancy rate and delivery.

DETAILED DESCRIPTION:
It has been common practice to cryopreserve surplus embryos achieved during IVF treatment or in other situation that embryos are to be preserved for other situations such as suspected ovarian hyper stimulation syndrome, fertility preservation or patient request.

Embryos are usually frozen on day 2, 3 or day 5-6 at the Blastocyst stage. At the time that thawing is planned, patients' cycle is synchronized and prepared either with hormonal treatment or at the natural cycle.

Not all embryos will always survive the thawing and sometimes they will all degenerate.

Embryos that survive the thawing procedure are assessed and replaced on the day of the thaw or left overnight for better selection and will be replaced only if they continue to divide in vitro.

The advantage of embryo transfer on the day of thaw is that embryo exposure in culture is shortened and embryo selection will be occurring in the womb. On the other hand, overnight incubation may avoid transferring embryos that potentially are not able to divide and are biologically not viable.

Although both attitudes are practiced in different IVF centers, at present there are no prospective randomized studies that have been conducted to advise which intervention is better in terms of pregnancy rates.

The purpose of the present study is to assess which technique will result in better pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* IVF patient who have thawed embryo transfer and can read understand and sigh on informed consent

Exclusion Criteria:

* IVF patient who have thawed embryo transfer and can not read understand and sigh on informed consent/ also those whos embryos will not survive freezing- thawing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 660 IVF patients. patients who are candidates for embryo cryopreservation cycle will be offered to participate in the present prospective randomized study.
  After detailed verbal and written explanation on the study protocol they will sign an informed consent and then randomized to 2 groups.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Pregnancy as measured by blood test for beta hCG | 12 days following embryos transfer
  as the usual routine, the women come on day 12 or 13 following embryo transfer to pur IVF unit to get blood teat for beta hCG. When the result show that the beta hCG is above 5 unit/liter we consider it as positive result and the patients is invited for additional blood test 2 days later/

SECONDARY OUTCOMES:
Delivery of baby | 9 mounth after embryos transfer
  We are routinely report to the Israeli ministry of health all the children who were born from our treatment. In this study we will calculate the number of children per thawed embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Dirnfeld, MD, Principal Investigator — Carmel Medical Center IVF Unit
Locations (1):
- Carmel Medical Center, Haifa, Israel

REFERENCES:
- [Background] Lahav-Baratz S, Koifman M, Shiloh H, Ishai D, Wiener-Megnazi Z, Dirnfeld M. Analyzing factors affecting the success rate of frozen-thawed embryos. J Assist Reprod Genet. 2003 Nov;20(11):444-8. doi: 10.1023/b:jarg.0000006705.46147.a2. PMID 14714822
- [Background] Lahav-Baratz S, Shiloh H, Koifman M, Kraiem Z, Wiener-Megnazi Z, Ishai D, Dirnfeld M. Early embryo-endometrial signaling modulates the regulation of matrix metalloproteinase-3. Fertil Steril. 2004 Oct;82 Suppl 3:1029-35. doi: 10.1016/j.fertnstert.2004.06.026. PMID 15474069